CLINICAL TRIAL: NCT04614051
Title: An Open Label, Single-center, Phase 1 Study to Evaluate the Safety of Cancer Immunotherapy With Autologous Dendritic Cells in Patients With Advanced or Recurrent Epithelial Ovarian Cancer
Brief Title: Safety Evaluation of Autologous Dendritic Cell Anticancer Immune Cell Therapy (Cellgram-DC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC-DC-02
Record Dates: First submitted 2020-10-22; First posted 2020-11-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellgram-DC (Experimental): Cellgram-DC is injected Subcutaneous injection near the upper arm lymph nodes
  Interventions: Biological: Cellgram-DC

INTERVENTIONS:
Biological: Cellgram-DC — Patients will receive 3 times every 2 weeks injection of Cellgram-DC(Autologous dendritic cell) subcutaneous injection near the upper arm lymph nodes
  Other Names: Autologous dendritic cell anticancer immune cell therapy for the treatment of ovarian cancer in patients with advanced or recurrent epithelial ovarian cancer

SUMMARY:
This Phase 1 study to evaluate the safety of cancer immunotherapy with autologous dendritic cells in patients with advanced or recurrent epithelial ovarian cancer

DETAILED DESCRIPTION:
To evaluate the safety of an autologous dendritic cell(DC) anticancer immune cell therapy (Cellgram-DC) for the treatment of advanced or recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 19 and under 80 years
2. Patients with Fédération Internationale de Gynécologie et d' Obstétrique(FIGO) stage III with histologically confirmed advanced or recurrent epithelial ovarian cancer (Serous, endometrioid, and mucinous only), fallopian tube cancer, and primary peritoneal cancer (residual tumor size <1cm)
3. Patients who have undergone tumor reduction or staging and complete or plan to complete platinum-based chemotherapy
4. In case of complete or partial response in primary or secondary chemotherapy
5. Whole body performance status: European Cooperative Oncology Group(ECOG) 0~1
6. Patients whose BRCA gene mutation test results can be confirmed
7. Patients whose life expectancy is at least 6 months or longer
8. Hb ≥ 8.0 g/dL, Absolute Neutrophil Count(ANC) ≥ 1,500/mm3, Platelets ≥ 100,000/mm3
9. Serum Creatinine ≤ 1.5 x Upper Limit of Normal(ULN) or Serum Creatinine> 1.5 x ULN and Calculated Creatinine Clearance> 30 mL/min
10. Total Bilirubin ≤ 1.5 x ULN or Direct bilirubin ≤ ULN, Aminotransferase (AST)/Alanine aminotransferase(ALT) <2.5 x ULN
11. Patients who did not receive surgery, radiation therapy, or immunotherapy within the last 6 weeks and recovered from side effects
12. Patients who agreed to use a medically recognized contraceptive method (diaphragm method used with spermicide, abstinence) during participation in the clinical trial (injection or implantable hormone therapy is not appropriate).
13. Patients who voluntarily participated in clinical trials and signed the Informed Contents Form (ICF)

Exclusion Criteria:

1. Patients with malignant tumors other than non-melanoma skin cancer in the past 3 years
2. Patients with brain metastases
3. Patients who previously received anti-tumor immunotherapy (anti-PD1, anti-PDL1 or anti-PDL2, etc.) or participated in immunotherapy-related clinical trials
4. Patients with active autoimmune diseases requiring systemic immunosuppression treatment (e.g., immunosuppressants such as cyclosporin A or azathioprine, or steroids for disease control)
5. Patients who use or plan to use Poly (ADP-ribose) polymerase (PARP) inhibitors due to the confirmed Breast Cancer Susceptibility Gene(BRCA) 1 or BRCA 2 mutation
6. Patients with medical conditions requiring continuous or intermittent administration of systemic steroids or immunosuppressants
7. Patients who received blood products (limited to whole blood products) within 4 weeks of screening criteria, or patients who received colony stimulating factors (Colony Stimulating Factor or recombinant Erythropoietin)
8. Patients with a history of organ or hematopoietic stem cell transplantation
9. Patients with acute or chronic infections requiring systemic treatment
10. Patients known to be infected with human immunodeficiency virus (HIV)/serum positive
11. Patients with active hepatitis A, B or C
12. Patients with untreated syphilis
13. Patients expected to need systemic chemotherapy, biotherapy, or immunotherapy for therapeutic purposes
14. Patients who received live virus vaccines (e.g. measles, mumps, rubella, chickenpox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), oral typhoid vaccine, Flu-Mist, etc.) within 30 days
15. Patients with a history of anaphylaxis to gentamicin
16. Pregnant or breastfeeding patients
17. Others, if the person in charge of the study determines that it is not suitable for the clinical trial

Ages: 19 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
The Measure CTCAE of Safety | -5, -3, 0, 2, 4, 8, 16 and 28 weeks
  The level of Adverse Event (AE) is described in accordance with the Common Terminology Criteria for Adverse Event (CTCAE) (Version 5.0).

SECONDARY OUTCOMES:
Immune response evaluation (INF-r) | 0, 2, 8, 16 and 28 weeks
  The tumor antigen-specific immune response induced after administration compared to before Investigational Product(IP) administration was confirmed by measuring changes in the secretion of cytokines (INF-r) in serum (ELISA).
Immune response evaluation (IL-12) | 0, 2, 8, 16 and 28 weeks
  The tumor antigen-specific immune response induced after administration compared to before Investigational Product(IP) administration was confirmed by measuring changes in the secretion of cytokines (IL-12) in serum (ELISA).
Measurement of changes in tumor marker test results (CA-125) | 0, 2, 4, 8, 16 and 28 weeks
  Changes in tumor marker test results (CA-125) are measured at each time point (V4, V5, V6, V7, V8) after administration compared to before (V3) Investigational Product(IP) administration.
Evaluation of solid tumor reflection at the time of follow-up observation | 8 and 28 weeks
  Responses of target/non-target lesions evaluated by the solid tumor reflection evaluation criteria (RECIST 1.1) at the time of follow-up (V6, V8)

CONTACTS AND LOCATIONS:
Overall Officials: Yongman Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea